CLINICAL TRIAL: NCT02774486
Title: Open-Label Clinical Investigation to Evaluate Efficacy and Safety of IQP-AK-102 on Appetite Reduction in Healthy Over- Weight Subjects
Brief Title: Efficacy and Safety of IQP-AK-102 in Reducing Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INQ/025115
Record Dates: First submitted 2016-03-22; First posted 2016-05-17 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Appetite Regulation; Appetite Suppression; Energy Intake

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IQP-AK-102 (Experimental): 2 capsules to be taken 3 times daily orally, 30 min before each main meal (breakfast, lunch, dinner) with 250 mL of water
  Interventions: Device: IQP-AK-102

INTERVENTIONS:
Device: IQP-AK-102 — IQP-AK-102 has been qualified as a medical device (CE certificate has been ob- tained), class IIb, according to MDD 93/42/EEC, annex IX, rule 5.

SUMMARY:
The primary cause of being overweight is an imbalance in calories consumed and energy expenditure. A surplus in energy intake might result in body fat deposition and thereby body weight gain. Therefore, food intake regulation is crucial to control the body weight gain.

Appetite regulation plays an important role in determining the food intake, which is a complex process influenced by the individual (physiology and psychology) and environment. Satiation (process that leads to the termination of eating) and satiety (decline in hunger, increase in fullness after a meal has finished) are the precursors of appetite regulation, which may be induced by various food components such as macronutrients, water, alcohol and non-digestible polysaccharides. High viscosity and swellable/bulking food components such as dietary fibre are expected to elicit stronger satiation/satiety than the macronutrients or clear liquid. Due to its unique physicochemical properties, dietary fibre has been recognized as potential ingredient that helps to enhance the sensation of satiety in the upper gut by increasing gastric distension and delaying gastric emptying, which subsequently reduces the food intake.

IQP-AK-102 comprises of a proprietary blend of dietary fibres known to promote a feeling a fullness. The objectives of this study are to evaluate the efficacy and safety of IQP-AK-102 on appetite reduction in overweight subjects during a 4-weeks interval.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, aged 18-65 years
2. BMI ≥25 and BMI <30 kg/m2
3. Generally in good health
4. Regular daily consumption of 3 main meals (breakfast, lunch, dinner)
5. Consistent regular physical activity (≤4 hours of strenuous sportive activity per week) AND willingness to maintain the same level of sport activity throughout the study
6. Commitment to avoid the use of other weight loss and/or management products / programmes during the study
7. Commitment to complete the subject diary correctly and to adhere to the lifestyle recommended for this study
8. Stable concomitant medications (if any)
9. Stable body weight for the last 3 months prior to V1 (less than 5% self-reported change)
10. Subject's agreement to comply with study procedures
11. Negative pregnancy testing (beta HCG-test in urine) at V1 in females of childbearing potential
12. Women of child-bearing potential: willingness to use reliable method of contraception during the study period

Exclusion Criteria:

1. Known sensitivity to the components of the investigational product
2. Bariatric surgery in the last 12 months prior to V1
3. Abdominal surgery within the last 6 months prior to V1
4. Presence of any active gastrointestinal disease incl. stenosis in the gastrointestinal tract
5. Malabsorption disorders
6. Pancreatitis
7. History of eating disorders like bulimia, anorexia nervosa, binge-eating (within the last 12 months prior to V1)
8. Lack of appetite for any (unknown) reason
9. Use of medications that could influence gastrointestinal functions such as antibiotics, laxatives, opioids, anticholinergics, anti-diarrheals 3 months prior to V1 and during the study
10. Use of medications that could influence body weight (e.g. antidepressants) in the last 3 months prior to V1 and during the study
11. Any medication or use of products for the treatment of obesity (e.g. fat binder, fat burner, satiety products etc.) or treatment that could influence food absorption, in last 3 months before V1 and during the study
12. Gluten allergy
13. History of abuse of drugs, alcohol or medication
14. Exceeding moderate alcohol consumption (≥21 units /week; 1 unit is equal 1⁄2 l of beer, or 200 ml of wine, or 50 ml hard liquor)
15. Smoking cessation within 6 months prior to V1 or during the study (regular smoking at the same level as prior to the study during the study is not an exclusion criteria)
16. Inability to comply with study procedures (e.g. due to language difficulties etc.)
17. Participation in similar studies or weight loss programs within the last 6 months prior to V1 and during the study
18. Participation in other clinical studies within the last 30 days prior to V1 and during the study
19. Clinically relevant deviations of laboratory values
20. Any other reason deemed suitable for exclusion, per investigator's judgement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-07-20 (Actual); Study Completion 2016-07-20 (Actual)

PRIMARY OUTCOMES:
Changes in appetite before and after breakfast 3 days a week (including one weekend day) using Haber Score (hunger, satiety) | 6 weeks
  - Comparison between week 2 and week 3 (first week of the IP intake) as well as comparison between week 2 and week 6 (last week of the IP intake)
Changes in appetite before and after breakfast 3 days a week (including one weekend day) using VAS (hunger, satiety, fullness, prospective food consumption). | 6 weeks
  - Comparison between week 2 and week 3 (first week of the IP intake) as well as comparison between week 2 and week 6 (last week of the IP intake)

SECONDARY OUTCOMES:
Changes in food intake using the subject diary | 6 weeks
  Measured on the same days as appetite assessment (for breakfast, lunch, dinner, in between meal/snacks), during the run-in phase (three days a week, both weeks) and treatment phase (at first week of the IP intake (week 3),and during the last week of the IP intake, just before the V3, also three days a week).
Changes in body weight using calibrated weighing scales (Tanita BC-420 SMA) | 6 weeks
  Body weight (kg) is measured in subjects wearing underwear and no shoes
Changes in BMI | 6 weeks
  BMI is calculated as body weight (kg)/(height [m])2
Changes in waist circumference | 6 weeks
  Waist circumference (cm) is measured at the level midway between the lateral lower rib margin and the iliac crest
Changes in hip circumference | 6 weeks
  Hip circumference (cm) is measured as the maximal circumference over the buttocks
Changes in body fat content using validated electronic weighing scales according to the Body composition analyser BC-420MA (a bio-impedance analysis (BIA)) | 6 weeks
  Measured as % and kg
Changes in fat-free mass using validated electronic weighing scales according to the Body composition analyser BC-420MA (a bio-impedance analysis (BIA)) | 6 weeks
  Measured as % and kg
Global evaluation of efficacy by subjects | 6 weeks
  The subjects will evaluate independently the efficacy of the IP (globally scaled evaluation with "very good", "good", "moderate" and "poor").
Global evaluation of efficacy by investigator | 6 weeks
  The investigators will evaluate independently the efficacy of the IP (globally scaled evaluation with "very good", "good", "moderate" and "poor").
Blood pressure | 6 weeks
  Measured using standard devices after an at least 5-minute rest
Pulse rate | 6 weeks
  Measured using standard devices after an at least 5-minute rest
Global evaluation of safety by subjects | 6 weeks
  The subjects will evaluate independently the tolerability of the IP (global scaled evaluation with "very good", "good", "moderate" and "poor").
Global evaluation of safety by investigator | 6 weeks
  The investigators will evaluate independently the tolerability of the IP (global scaled evaluation with "very good", "good", "moderate" and "poor").

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Uebelhack, MD, PhD, Principal Investigator — analyze & realize GmbH
Locations (1):
- Barbara Grube, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No